CLINICAL TRIAL: NCT06982157
Title: A Comparison Between Vaginal Sacrospinous Ligament Fixation and Laparoscopic Uterosacral Ligament Suspension as a Uterine Preserving Surgery for Pelvic Organ Prolapse
Acronym: POP-Q USS USLS
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: 0111-20-HYMC
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Pelvic Organ Prolapse (POP); Pelvic Organ Prolapse Vaginal Surgery; Hysterectomy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaginal sacrospinous ligament fixation: Vaginal sacrospinous ligament fixation
- laparoscopic uterosacral ligament suspension: laparoscopic uterosacral ligament suspension

SUMMARY:
The investigators present a literature review evaluating the current place of sacrospinous hysteropexy in the surgical management of pelvic organ prolapse. Additionally, to assess the efficacy of the procedure, the investigators performed a meta-analysis comparing sacrospinous hysteropexy with vaginal hysterectomy and repair in terms of anatomical outcomes, complications, and repeat surgery rates.

Vaginal sacrospinous ligament fixation is associated with less anatomic recurrent prolapse and prolapse related symptoms compared with laparoscopic uterosacral ligament suspension in women desiring uterine preservation Hypothesis: Vaginal SSF and lap USLS may have comparable anatomic outcomes in repair of mild to mod uterine prolapse but LUSLS may be associated with longer OT while SSF with more post-op pelvic pain and a higher rate of future prolapse at the ant. Compartment.

Objective: In this study we aim to evaluate the risk of anatomic and symptomatic POP after vaginal sacrospinous ligament fixation and laparoscopic uterosacral ligament suspension among patients who underwent pelvic organ prolapse repair at a single university-affiliated maternity hospital, by comparing the clinical (symptoms - questionnaires) and anatomical (POP Q) outcomes between the two techniques 6, 12, 18, and 24 months following surgery, and therefore establishing personalized approach relying on pre-op parameters.

Specific Aims

* Specific aim 1: Evaluate the efficacy and safety of vaginal sacrospinous ligament fixation and laparoscopic uterosacral ligament suspension among patients who underwent pelvic organ prolapse repair at HY medical center.
* Specific aim 2: Compare the clinical (symptoms - questionnaires) and anatomical (POP Q) outcomes between the two techniques 6, 12, 18, and 24 months following surgery.
* Specific aim 3: Determine the patient characteristics that might delineate which surgery is appropriate for the given group.

DETAILED DESCRIPTION:
Vaginal hysterectomy, with or without repair, is the most common procedure performed for apical prolapse. The underlying etiology of apical prolapse is a weakness in the supports of the uterus and upper vagina. There is a growing body of evidence to suggest that uterine preserving procedures for treatment of prolapse are effective and safe. Vaginal sacrospinous hysteropexy is a relatively simple procedure which can be carried out by the generalist gynecologist who performs vaginal repairs.

Sacrospinous hysteropexy is a safe and effective procedure for pelvic organ prolapse and has comparable outcomes to vaginal hysterectomy with repair.

Hysterectomy with laparoscopic uterosacral colpopexy has been shown to produce better objective success rates than laparoscopic uterosacral hysteropexy; however, repeat operation rates are not significantly different.

The surgical management of multi-compartment prolapse is challenging and often requires a combination of techniques.

ELIGIBILITY:
Inclusion Criteria:

* From the general Urogynecological cohort who underwent vaginal sacrospinous suspension and laparoscopic uterosacral Sacrospinous ligament fixation at Hillel Yaffe Hospital.

Exclusion Criteria:

* None

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women who underwent vaginal sacrospinous suspension and laparoscopic uterosacral Sacrospinous ligament fixation
Study Population: Women who underwent vaginal sacrospinous suspension and laparoscopic uterosacral Sacrospinous ligament fixation
Sampling Method: Non-Probability Sample
Enrollment: 111 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Risks of anatomic POP after vaginal sacrospinous ligament fixation and laparoscopic uterosacral ligament suspension | 2 years
  Evaluate the risk of anatomic POP after vaginal sacrospinous ligament fixation and laparoscopic uterosacral ligament suspension among patients who underwent pelvic organ prolapse repair.
  The evaluation will be carried out by comparing the clinical (symptoms - questionnaires) and anatomical (POP Q) outcomes between the two techniques 6, 12, 18, and 24 months following surgery, and therefore establishing personalized approach relying on pre-op parameters.
Risks of symptomatic POP after vaginal sacrospinous ligament fixation and laparoscopic uterosacral ligament suspension | 2 years
  Evaluate the risk of symptomatic POP after vaginal sacrospinous ligament fixation and laparoscopic uterosacral ligament suspension among patients who underwent pelvic organ prolapse repair. The evaluation will be carried out by comparing the clinical (symptoms - questionnaires) and anatomical (POP Q) outcomes between the two techniques 6, 12, 18, and 24 months following surgery, and therefore establishing personalized approach relying on pre-op parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Jonia Alsheik, Dr, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hille Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: Undecided